CLINICAL TRIAL: NCT00000228
Title: Buprenorphine Detox With Two Types of Treatment. BBD I
Brief Title: Buprenorphine Detox With Two Types of Treatment. BBD I - 10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Purpose: Treatment
Other Study IDs: NIDA-06969-10; R01-06969-10
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 1996-07

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to compare overall treatment outcome between behavioral versus standard treatment types.

ELIGIBILITY:
Please contact site for information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1994-08

PRIMARY OUTCOMES:
Drug use
Retention
Weeks abstinent
Weeks continuous abstinence
Overall treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States

REFERENCES:
- [Background] Bickel WK, Amass L, Higgins ST, Badger GJ, Esch RA. Effects of adding behavioral treatment to opioid detoxification with buprenorphine. J Consult Clin Psychol. 1997 Oct;65(5):803-10. doi: 10.1037//0022-006x.65.5.803. PMID 9337499